CLINICAL TRIAL: NCT00419991
Title: An Open-Label Noncomparative, Multicenter, Clinical Trail Measuring Time Related Clinical Response Factors in Relation to Time to Bacterial Eradication With Tigecycline Treatment in Patients With Catheter Infection
Brief Title: Open Label Non-comparative Clinical Trial of Tigecycline in Patients With Catheter Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CPL Associates (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Jerome Schentag, Pharm.D., CPL Associates, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPLA-6625
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Staphylococcal Infections
Keywords: Tigecycline; Staphylococcal Infections; Catheter
MeSH Terms: conditions — Staphylococcal Infections | interventions — Tigecycline

ARMS (1):
- 1 Tigecycline (No Intervention)
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — All patients will receive tigecycline infusions approximately every 12 or 24 hours. The usual regimen of tigecycline is (an initial intravenous (IV) dose of 100 mg followed by 50 mg approximately every 12 hours). Patients with severe hepatic dysfunction may, at the investigator's discretion with CPL Associates approval (call enrollment hotline) may be given a total daily dose of 50 mg (one 50 mg dose or 25 mg approximately every 12 hours). Tigecycline infusions will be administered over approximately 30 minutes in 100 mL of normal saline.

SUMMARY:
Tigecycline is being developed as an agent that overcomes tetracycline-resistance mechanisms and provides activity against emerging multi-drug resistant pathogens. The purpose of this protocol is to determine the linkage between time related clinical measures of infection response and time to bacterial eradication in patients with intravascular catheter infections caused by Staphylococcus epidermidis and other coagulase negative staphylococci.

DETAILED DESCRIPTION:
Tigecycline, a glycylcycline antibiotic and an analog of the tetracycline minocycline, demonstrates a broad spectrum of antibacterial activity by inhibiting multiply resistant gram-positive, gram-negative, anaerobic, and "atypical" bacteria. It is being developed as an agent that overcomes tetracycline-resistance mechanisms and provides activity against emerging multi-drug resistant pathogens. These attributes may provide clinicians with a valuable therapeutic alternative. The purpose of this protocol is to determine the linkage between time related clinical measures of infection response and time to bacterial eradication in patients with intravascular catheter infections caused by Staphylococcus epidermidis and other coagulase negative staphylococci. The study is being conducted in two phases. The first treats patients who have removal of the catheter at the time of treatment, and the second treats patients who have the catheter remaining in situ during tigecycline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18-85 years of age and a weight of > 45 kilograms.
* Patients with intravascular catheters and a blood culture that is positive for gram-positive cocci in clusters. Patients will be subsequently excluded from the study analysis if they do not have a culture-positive infection with S. epidermidis or other coagulase negative staphylococci, expected to be susceptible to tigecycline.
* Patients in whom the bacteremia can be cultured daily by the site investigator.
* Patients who have failed other available antibiotic therapies may be enrolled with positive blood cultures and organism susceptibility to tigecycline.

Exclusion Criteria:

* Patients that cannot be cultured daily by the site investigator.
* Intravascular catheter infections known to be caused by bacteria other than a coagulase negative staphylococci, for example, Staphylococcus aureus.
* Any patient who has received more than 24 hrs of vancomycin.
* Any patient who has received any antibiotic active against S. epidermidis other than vancomycin.
* Patients who are moribund with an expected survival of less than 2 weeks.
* Patients who are neutropenic (ANC <500) at the time of bacteremia
* Patients who have been designated as "Do Not Resuscitate", unless it is anticipated within a reasonable degree of medical certainty that they can achieve benefit from tigecycline therapy.
* Known or suspected hypersensitivity to tigecycline, tetracyclines, or other compounds related to this class of antibacterial agents.
* Pregnant women or nursing mothers.
* Female patients of childbearing potential who do not agree to use a medically acceptable method of contraception throughout the duration of the study and for at least 1 month after the last dose of tigecycline.
* Patients with suspected or proven endocarditis or osteomyelitis
* Patients with suspected or proven mycobacterial infections

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to bacterial eradication | 7-14 days

SECONDARY OUTCOMES:
Safety and Efficacy of Tigecycline in patients with intravascular catheter infections | 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G Maki, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - CPL Associates Investigational Site, Huntsville, Alabama
  - CPL Associates Investigational Site, Marietta, Georgia
  - CPL Associates Investigational Site, Cumberland, Maryland

REFERENCES:
- [Background] Schnappinger D, Hillen W. Tetracyclines: antibiotic action, uptake, and resistance mechanisms. Arch Microbiol. 1996 Jun;165(6):359-69. doi: 10.1007/s002030050339. PMID 8661929
- [Background] Gales AC, Jones RN. Antimicrobial activity and spectrum of the new glycylcycline, GAR-936 tested against 1,203 recent clinical bacterial isolates. Diagn Microbiol Infect Dis. 2000 Jan;36(1):19-36. doi: 10.1016/s0732-8893(99)00092-9. PMID 10744364
- [Background] Meinl B, Hyatt JM, Forrest A, Chodosh S, Schentag JJ. Pharmacokinetic/pharmacodynamic predictors of time to clinical resolution in patients with acute bacterial exacerbations of chronic bronchitis treated with a fluoroquinolone. Int J Antimicrob Agents. 2000 Nov;16(3):273-80. doi: 10.1016/s0924-8579(00)00253-3. PMID 11091047
- [Background] Ambrose PG, Anon JB, Owen JS, Van Wart S, McPhee ME, Bhavnani SM, Piedmonte M, Jones RN. Use of pharmacodynamic end points in the evaluation of gatifloxacin for the treatment of acute maxillary sinusitis. Clin Infect Dis. 2004 Jun 1;38(11):1513-20. doi: 10.1086/420739. Epub 2004 May 12. PMID 15156435
- See also: CPL Associates Website — http://www.cplassociates.com